CLINICAL TRIAL: NCT01863225
Title: A Phase 2 Multiple-Dose Study to Characterize the Pharmacokinetics of RVX000222 Capsule Formulation in Combination With Either Atorvastatin or Rosuvastatin in Patients With Dyslipidemia
Brief Title: Characterization of Multi-dose RVX000222 in Combination With Statin Treatment in Dyslipidemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Resverlogix Corp (Industry)
Collaborators: South Australian Health and Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RVX222-CS-009
Record Dates: First submitted 2013-05-16; First posted 2013-05-27 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Dyslipidemia; Coronary Artery Disease
MeSH Terms: conditions — Dyslipidemias; Coronary Artery Disease | interventions — apabetalone; Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): RVX000222 200 mg (100 mg b.i.d.) + Atorvastatin 40 mg
  Interventions: Drug: RVX000222; Drug: Atorvastatin
- Group B (Experimental): RVX000222 200 mg (100 mg b.i.d.) + Rosuvastatin 20 mg
  Interventions: Drug: RVX000222; Drug: Rosuvastatin
- Group C (Experimental): RVX000222 200 mg (100 mg b.i.d.) + Atorvastatin 80 mg
  Interventions: Drug: RVX000222; Drug: Atorvastatin
- Group D (Experimental): RVX000222 200 mg (100 mg b.i.d.) + Rosuvastatin 40 mg
  Interventions: Drug: RVX000222; Drug: Rosuvastatin

INTERVENTIONS:
Drug: RVX000222 — capsule, 200 mg, administer with food, 100 mg twice daily 10-12 hrs apart, 14-days
  Other Names: RVX-208
Drug: Rosuvastatin — 20 mg daily, 28-42 days
  Arms: Group B
Drug: Atorvastatin — 40 mg daily, 28-42 days
  Arms: Group A
Drug: Rosuvastatin — 40 mg daily, 28-42 days
  Arms: Group D
Drug: Atorvastatin — 80 mg daily, 28-42 days
  Arms: Group C

SUMMARY:
This study is designed to characterize the pharmacokinetics of multi-dose RVX000222 and atorvastatin and rosuvastatin when either statin is administered in combination with RVX000222 in subjects with dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 18 to ≤ 65 years of age with or without documented coronary artery disease.
* Taking statin therapy for at least 30 days prior to Screening (Visit 1).
* In the opinion of the investigator, patient currently on statin therapy other than atorvastatin 40 mg or rosuvastatin 20 mg or atorvastatin 80 mg or rosuvastatin 40 mg who could be switched to one of these regimens at Visit 1 for the duration of the study.

Exclusion Criteria:

* Clinically significant heart disease which will require coronary bypass, PCI, cardiac transplantation, surgical repair and/or replacement during the course of the study.
* Coronary artery bypass graft (CABG) procedure within the past 90 days.
* Have a body mass index (BMI) greater than 36 kg/m2.
* Patients of East Asian descent (due to pharmacological food effect noted for rosuvastatin).
* Previous or current diagnosis of severe heart failure (NYHA Class III-IV) or a documented left ventricular ejection fraction (LVEF) of < 25% as determined by contrast left ventriculography, radionuclide ventriculography or echocardiography. The absence of an LVEF measurement in a patient without a previous or current diagnosis of heart failure does not prohibit entry into the study.
* Patients with evidence of cardiac electrophysiologic instability including a history of uncontrolled ventricular arrhythmias, uncontrolled atrial fibrillation/flutter or uncontrolled supraventricular tachycardias with a ventricular response heart rate of > 100 beats per minute at rest within 4 weeks prior to Visit 1.
* Evidence of renal impairment
* Have hypertension that is uncontrolled defined as 2 consecutive measurements of sitting blood pressure of systolic >160 mmHg or diastolic > 95 mmHg at Visit 1.
* Women of child-bearing potential who do not agree to use two reliable methods of birth control during the study and for one month following the last dose of study drug, or pregnant or nursing (lactating) women. Where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive ß-hCG laboratory test (≥ 5 IU/L) at the time of enrollment. Where women of child-bearing potential are defined as women not surgically sterilized and between menarche and 1 year post menopause, and a reliable method of birth control includes use of oral contraceptives or levonorgestrel; or a reliable barrier method of birth control (diaphragms; cervical caps; condoms; intrauterine devices; partner with vasectomy; or abstinence).
* Current or recent (within 12 month prior to Visit 1) treatment with immunosuppressants (e.g., Cyclosporine).
* Triglycerides > 4.5 mmol/L at screening Visit 1.
* Use of fibrates of any dose or niacin/nicotinic acid 250 mg or more within 90 days prior to Visit 1
* Any medical or surgical condition which might significantly alter the absorption, distribution, metabolism or excretion of medication including, but not limited to any of the following: cholecystitis, Crohn's disease, ulcerative colitis, or any gastric bypass alteration.
* Evidence of hepatic disease
* A total bilirubin that is > ULN by local laboratory at screening, Visit 1
* History of malignancy of any organ system, treated or untreated, within the past 5 years of Visit 1 whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.
* History or evidence of drug or alcohol abuse within 12 months of Visit 1.
* Current dependence on nicotine containing products.
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study.
* Use of any HIV and/or chemotherapy drugs, and/or antibiotics within 30 days or 5 half-lives of Visit 2, whichever is longer.
* Use of other investigational drugs and devices at the time of enrollment, or within 30 days or 5 half-lives of Visit 2, whichever is longer.
* History of noncompliance to medical regimens or unwillingness to comply with the study protocol.
* Any condition that in the opinion of the investigator would confound the evaluation and interpretation of efficacy and/or safety data.
* Persons directly involved in the execution of this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Characterization of the pharmacokinetics of RVX000222 capsule formulation in combination with either atorvastatin or rosuvastatin in patients with dyslipidemia. | 14 days
  The plasma concentration-time profile of RVX000222 capsule formulation and its metabolites on Days 1 and 14 of 200 mg daily RVX000222 in combination with either atorvastatin or rosuvastatin, including pharmacokinetic parameters Cmax, Tmax, Cmin, AUC0-12, AUC12-24, AUC0 24, and metabolite ratio.

SECONDARY OUTCOMES:
Characterization of the pharmacokinetics of atorvastatin and rosuvastatin when either is administered in combination with RVX000222 capsule formulation to patients with dyslipidemia. | 14 days
  The plasma concentration-time profile of either atorvastatin and metabolites or rosuvastatin and metabolites on Days -1 and 14 of 200 mg daily RVX000222 in combination with the statin, including pharmacokinetic parameters Cmax, Tmax, Cmin, AUC0-12, AUC12-24, AUC0 24, and metabolite ratio.
Evaluation of safety and tolerability of RVX000222 capsule formulation administered in combination with stable doses of either atorvastatin or rosuvastatin in patients with dyslipidemia. | 14
  Adverse events, serious adverse events, vital signs, clinical chemistry and haematological variables will be collected and summarized across treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Sepehr Shakib, Principal Investigator — Royal Adelaide Hospital
Locations (1):
- Royal Adelaide Hospital / CMAX, Adelaide, South Australia, Australia